CLINICAL TRIAL: NCT03254927
Title: A Phase 2, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of CDX-3379 in Combination With Cetuximab in Patients With Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of CDX-3379 and Cetuximab and in Patients With Advanced Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on emerging risk-benefit profile
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX3379-04
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Advanced Head and Neck Squamous Cell Carcinoma
Keywords: Erbitux; Cetuximab; Oral Cancer; Oropharyngeal cancer; Laryngeal cancer; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDX-3379 and cetuximab (Experimental): During the treatment phase of the study, eligible patients will receive assigned treatments in 3 week cycles until progression.
  Interventions: Drug: CDX-3379 and cetuximab

INTERVENTIONS:
Drug: CDX-3379 and cetuximab — Dose: 12 mg/kg CDX-3379 once every 3 weeks in combination with 400 mg/m2 cetuximab on the first day followed by weekly doses of 250 mg/m2 cetuximab.

SUMMARY:
This is a study to determine the clinical benefit (how well the drug works), safety and tolerability of combining CDX-3379 and cetuximab. The study will enroll patients with advanced head and neck squamous cell carcinoma who have previously received cetuximab and progressed.

DETAILED DESCRIPTION:
CDX-3379 is a fully human monoclonal antibody that binds to a molecule called human epidermal growth factor receptor 3 (HER3 or ErbB3) found on certain cells and may act to promote anti-tumor effects.

Cetuximab is a human monoclonal antibody that blocks EGFR, a protein receptor that regulates cell growth.

This study will evaluate the safety, tolerability and efficacy of CDX-3379 in combination with cetuximab in patients with advanced head and neck squamous cell carcinoma who have previously received cetuximab and progressed.

Eligible patients that enroll in the study will be given the dose of 12 mg/kg CDX-3379 once every 3 weeks in combination with 400 mg/m2 cetuximab on the first day followed by weekly doses of 250 mg/m2 cetuximab.

Up to 45 patients will be enrolled. All patients enrolled in the study will be closely monitored to determine if there is a response to the treatment as well as for any side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed head and neck squamous cell carcinoma.
2. Human papilloma virus (HPV) negative tumor.
3. Prior treatment with a check-point inhibitor targeting PD-1, unless not a candidate.
4. Prior treatment with cetuximab with tumor progression during or within 6 months after completing treatment.
5. Measurable disease.
6. Life expectancy ≥ 12 weeks.
7. If of childbearing potential (male or female), agrees to practice an effective form of contraception during study treatment and for at least 6 months following last treatment.
8. Willingness to undergo a tumor biopsy prior to starting treatment (or if biopsy is not feasible, provide archival tissue).

Exclusion Criteria:

1. Previous treatment with CDX-3379 or other anti-ErbB3 targeted agents.
2. Nasal, paranasal sinus, or nasopharyngeal carcinoma, aside from WHO Type I and II (keratinizing, non-EBV positive) nasopharyngeal carcinoma which will be allowed.
3. Major surgery within 4 weeks prior to first dose of study treatment.
4. Chemotherapy within 21 days or at least 5 half-lives (whichever is shorter) prior to first dose of study treatment.
5. Monoclonal based therapies within 4 weeks (excluding cetuximab) and all other immunotherapy within 2 weeks prior to first dose of study treatment.
6. Other prior malignancy, active within 3 years, except for localized prostate cancer, cervical carcinoma in situ, non-melanomatous carcinoma of the skin, stage 1 differentiated thyroid cancer or ductal carcinoma in situ of the breast.
7. Active, untreated central nervous system metastases.
8. Active autoimmune disease or documented history of autoimmune disease.
9. Significant cardiovascular disease including CHF or poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Rush University Medical center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania Hospital, Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Duvvuri U, George J, Kim S, Alvarado D, Neumeister VM, Chenna A, Gedrich R, Hawthorne T, LaVallee T, Grandis JR, Bauman JE. Molecular and Clinical Activity of CDX-3379, an Anti-ErbB3 Monoclonal Antibody, in Head and Neck Squamous Cell Carcinoma Patients. Clin Cancer Res. 2019 Oct 1;25(19):5752-5758. doi: 10.1158/1078-0432.CCR-18-3453. Epub 2019 Jul 15. PMID 31308059

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CDX-3379 and Cetuximab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CDX-3379 and Cetuximab
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 62 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30
Site of Primary Tumor [Count of Participants; unit: Participants]
  Pharynx/Oropharynx | 12
  Oral Cavity | 11
  Larynx | 4
  Other | 3
Duration of Metastatic Disease [Mean (Full Range); unit: years] | 2.2 [1 to 17]
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status as published in Am. J. Clin. Oncol (Oken, et al. 1982) 0 = Fully active, able to carry on all pre-disease performance without restriction.
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG 0 | 4
    ECOG 1 | 26

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The percentage of patients who achieve a complete response or partial response per Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST version 1.1), Complete Response (CR) = disappearance of all target lesions and non-target lesions, Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions with no progression in non-target lesions and no new lesions.
Time Frame: The proportion of evaluable patients who achieve a best overall response of complete or partial response according to RECIST 1.1 assessed up to 24 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CDX-3379 and Cetuximab
Number analyzed (Participants) | 30
percentage of participants | 7 [0.8 to 22.1]

2. Secondary Outcome: Clinical Benefit Response (CBR)
Description: The percentage of patients who achieve best response of confirmed CR or PR, or stable disease (SD) for at least 12 weeks
Time Frame: Every 8 weeks, starting with first dose until disease progression, assessed up to approximately 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CDX-3379 and Cetuximab
Number analyzed (Participants) | 30
percentage of participants | 40 [22.7 to 59.4]

3. Secondary Outcome: Duration of Response (DOR)
Description: The interval from which measurement criteria are first met for Complete Response (CR) or Partial Response (PR) until the first date that progressive disease is objectively documented
Time Frame: First occurrence of a documented objective response to disease progression or death (up to approximately 2 years)
Measure: Number; unit: months
Arm/Group | CDX-3379 and Cetuximab
Number analyzed (Participants) | 30
months | NA — 30 patients were treated, 2 patients achieved objective response. The duration of response was 5 months and 18.7 months for the 2 patients who achieved objective response.

4. Secondary Outcome: Progression-free Survival (PFS)
Description: The time from start of study drug to time of progression or death, whichever occurs first
Time Frame: From first dose to the first occurrence of disease progression or death due to any cause (up to approximately 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CDX-3379 and Cetuximab
Number analyzed (Participants) | 30
months | 2.2 [1.3 to 3.6]

5. Secondary Outcome: Overall Survival (OS)
Description: The time from start of study drug to death
Time Frame: The time from start of study drug to death from any cause (up to approximately 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CDX-3379 and Cetuximab
Number analyzed (Participants) | 30
months | 6.6 [2.7 to 7.5]

6. Secondary Outcome: Incidence of Adverse Events [Safety and Tolerability]
Description: Safety and tolerability of CDX-3379 in combination with cetuximab as determined by incidence and severity of adverse events. Percentage of patients reporting one or more adverse events.
Time Frame: Following at least one dose of study treatment through 30 days after last dose of CDX-3379.
Measure: Count of Participants; unit: Participants
Arm/Group | CDX-3379 and Cetuximab
Number analyzed (Participants) | 30
Participants | 30

7. Secondary Outcome: Tumor DNA Biomarkers.
Description: Tumor DNA biomarkers will be evaluated and assessed for correlation with clinical efficacy. Objective response rate for subset of patients with FAT1 positive tumor is reported.
Time Frame: Tumor tissue is obtained during screening window via single biopsy procedure.
Population: patients with FAT1 positive tumors
Measure: Count of Participants; unit: Participants
Arm/Group | CDX-3379 and Cetuximab
Number analyzed (Participants) | 10
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from initiation of treatment until 30 days after discontinuing treatment or initiation of new anti-cancer medication.
Arm/Group | CDX-3379 and Cetuximab
All-Cause Mortality (participants affected / at risk) | 26/30
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CDX-3379 and Cetuximab (N=30)
Pneumonia (Infections and infestations) | 3
Lung abscess (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Mucosal inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CDX-3379 and Cetuximab (N=30)
Diarrhoea (Gastrointestinal disorders) | 24
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 16
Hypokalaemia (Metabolism and nutrition disorders) | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 6
Malnutrition (Metabolism and nutrition disorders) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hypernatraemia (Metabolism and nutrition disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 17
Dry skin (Skin and subcutaneous tissue disorders) | 8
Skin induration (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Pruritis (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 11
Asthenia (General disorders) | 2
Chills (General disorders) | 5
Thirst (General disorders) | 2
Face oedema (General disorders) | 3
Catheter site pain (General disorders) | 2
Weight decreased (Investigations) | 10
Blood creatinine increased (Investigations) | 6
Blood lactate dehydrogenase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 2
Amylase increased (Investigations) | 3
Lipase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 2
International normalised ratio increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Dizziness (Nervous system disorders) | 6
Presyncope (Nervous system disorders) | 3
Headache (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 3
Paronychia (Infections and infestations) | 4
Skin infection (Infections and infestations) | 3
Fungal skin infection (Infections and infestations) | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 2
Skin laceration (Injury, poisoning and procedural complications) | 2
Anaemia (Blood and lymphatic system disorders) | 7
Blepharitis (Eye disorders) | 2
Vision blurred (Eye disorders) | 2
Proteinuria (Renal and urinary disorders) | 5
Hypotension (Vascular disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Confusional state (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Agitation (Psychiatric disorders) | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Fall (Injury, poisoning and procedural complications) | 3

LIMITATIONS AND CAVEATS:
Study was terminated early due to unfavorable risk/benefit profile.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT03254927/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT03254927/SAP_001.pdf